CLINICAL TRIAL: NCT02518282
Title: High-sensitivity Troponin T in Acute Myocardial Infarction in Patients Undergoing Cardiac Valvular Surgery
Brief Title: High-sensitivity Troponin T in Acute Myocardial Infarction After Cardiac Valvular Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Valladolid (Other)
Responsible Party: Principal Investigator, Héctor Cubero Gallego, MD, University of Valladolid
Other Study IDs: PI 15-223 CINV 15-01
Record Dates: First submitted 2015-08-04; First posted 2015-08-07 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Acute Myocardial Infarction; Disorder; Heart, Functional, Postoperative, Cardiac Surgery; Myocardial Infarction; Heart Valve Diseases
Keywords: high-sensitivity troponin T; Acute myocardial infarction; Heart valvular surgery; Cardiac surgery
MeSH Terms: conditions — Myocardial Infarction; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Serum levels of high-sensitivity troponin T — Serum levels of hs-cTn will be measured before surgery, upon arrival at the ICU, as well as every 6 hours for 24 hours, then every 8 hours the following 24 hours and a last blood sample will be taken 72 hours after surgery.
Other: Twelve-lead ECGs — Twelve-lead ECGs obtained the day prior to heart valvular surgery, immediately upon arrival at the ICU, and then 24, 48 and 72 hours post-surgery will be reviewed by a cardiologist to evidence signs of MI.
Other: Transthoracic echocardiography (TTE) — A TTE will be also performed by a cardiologist after cardiac valvular surgery to determine the ejection fraction of left ventricle and the occurrence of a new regional wall motion abnormality. This TTE will be compared, by the same cardiologist, with a TTE performed before cardiac valvular surgery.

SUMMARY:
A measurable degree of heart muscle tissue injury is expected in patients undergoing heart valvular surgery. The level of this injury can be measured by cardiac biomarkers in blood samples. Those biomarkers are used to diagnose an acute myocardial infarction.

Postoperative myocardial infarction (MI) is a frequent and important complication after cardiac surgery with high morbidity and mortality. Therefore it is very important to recognize any cardiac event in patients who undergo cardiac surgery. Different diagnostic tools can be used to the diagnosis of acute myocardial infarction; however few is known about the value of high-sensitivity cardiac troponin T (hs-cTn) to diagnose a MI after heart valvular surgery.

The aim of this study is to determine the upper reference limit of high-sensitivity troponin T concentration to consider the diagnosis of acute myocardial infarction in patients undergoing heart valvular surgery.

DETAILED DESCRIPTION:
This is a longitudinal prospective observational cohort mono centre study. Hs-cTn will be measured at different point of times in adult patients undergoing heart valvular surgery with cardiopulmonary bypass (CPB) and without recent medical history of ischemic heart disease.

The study is conducted at the University Clinical Hospital of Valladolid, Spain. The Cardiac Surgery department annually performs approximately 550 cardiac surgeries with CPB in adult patients (approximately 300 heart valvular surgeries). Two operating rooms are routinely used. There is an intensive care unit (ICU) with 10 beds dedicated exclusively to the postoperative care of patients who undergo cardiac surgery.The hospital's research commission approved the study. All patients, preoperatively, provided informed written consent both for their heart surgery and for their participation in the study.

Serum levels of hs-cTn will be measured before cardiac surgery, upon arrival at the ICU, as well as every 6 hours for 24 hours, then every 8 hours the following 24 hours and a last blood sample will be taken 72 hours after cardiac surgery. Samples are analysed at the department of Clinical Biochemistry of our hospital.

Twelve-lead electrocardiograms (ECGs) obtained the day prior to heart valvular surgery, immediately upon arrival at the ICU, and then 24, 48 and 72 hours post-surgery will be reviewed by a cardiologist to evidence signs of myocardial infarction (MI). All cardiac events will be noted as The Third Global MI Task Force definition of MI describes.

A transthoracic echocardiography (TTE) will be also performed by a cardiologist after cardiac valvular surgery to determine the ejection fraction of left ventricle and the occurrence of a new regional wall motion abnormality. This TTE will be compared, by the same cardiologist, with a TTE performed before cardiac valvular surgery.

The principal investigator will supervise data handling.

ELIGIBILITY:
Inclusion Criteria:

* Each participant must be older than 18 years.
* Undergoing cardiac valvular surgery.
* No recent clinical history of ischemic heart disease.
* Each participant must voluntarily give his written informed consent.

Exclusion Criteria:

* Patients undergoing coronary bypass artery grafting (CABG).
* Patients with severe or end-stage renal insufficiency.
* Insertion of assist devices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (over 18 years old) undergoing heart valvular surgery with CPB.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-04 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Determination of upper reference limit (URL) of high-sensitivity troponin T that strongly suggests substantial myocardial damage and necrosis. | Every 6 postoperative hours for the first 24 hours, then every 8 hours the following 24 hours and a last sample will be taken 72 hours after heart valvular surgery.
  Postoperative MI remains a frequent complication after cardiac surgery with high morbidity and mortality. In 2012 the Third Global MI Task Force presented the third universal definition of MI implying that MI associated with coronary artery bypass grafting (CABG) is arbitrarily defined by elevation of cardiac biomarkers values over 10 x 99th percentile URL in patients with normal baseline cTn values. In addition with either: a) new pathological Q waves or new left bundle branch block (LBBB), or b) angiographic documented new graft or new native coronary artery occlusion, or c) imaging evidence of new loss of viable myocardium or new regional wall motion abnormality. Few is known about the established threshold values for hs-cTn after heart valvular surgery.

SECONDARY OUTCOMES:
High-sensitivity troponin T concentration changes over time in patients undergoing heart valvular surgery | From 8 hours preoperatively to 72 hours postoperatively
  Serum levels of hs-cTn will be measured before cardiac surgery, upon arrival at the ICU, as well as every 6 hours for 24 hours, then every 8 hours the following 24 hours and a last blood sample will be taken 72 hours after heart valvular surgery.
Number of patients with complications after heart valvular surgery. | After cardiac valvular surgery to 72 hours post-surgery.
  To determine the number of patients with complications after heart valvular surgery and to determine which are the most frequent complications in patients undergoing cardiac valvular surgery.

OTHER OUTCOMES:
Twelve-lead ECGs. | The day prior to cardiac surgery, immediately upon arrival at the ICU, and then 24, 48 and 72 hours post-surgery.
  Twelve-lead ECGs will be reviewed by a cardiologist to evidence signs of postoperative MI.
Transthoracic Echocardiography (TTE). | Before heart valvular surgery and after heart valvular surgery.
  A TTE will be performed after heart valvular surgery to evidence a new regional wall motion abnormality. This TTE will be compared with a TTE performed before surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Héctor Cubero Gallego, MD, Principal Investigator — University Clinical Hospital of Valladolid; Eduardo Tamayo Gómez, MD, PhD, Study Chair — University Clinical Hospital of Valladolid; José Alberto San Román Calvar, MD, PhD, Study Chair — University Clinical Hospital of Valladolid; José Ignacio Gómez Herreras, MD, PhD, Study Chair — University Clinical Hospital of Valladolid
Locations (1):
- University Clinical Hospital of Valladolid, Valladolid, Spain, Spain

REFERENCES:
- [Result] Thygesen K, Mair J, Katus H, Plebani M, Venge P, Collinson P, Lindahl B, Giannitsis E, Hasin Y, Galvani M, Tubaro M, Alpert JS, Biasucci LM, Koenig W, Mueller C, Huber K, Hamm C, Jaffe AS; Study Group on Biomarkers in Cardiology of the ESC Working Group on Acute Cardiac Care. Recommendations for the use of cardiac troponin measurement in acute cardiac care. Eur Heart J. 2010 Sep;31(18):2197-204. doi: 10.1093/eurheartj/ehq251. Epub 2010 Aug 3. PMID 20685679
- [Result] Morrow DA, Cannon CP, Jesse RL, Newby LK, Ravkilde J, Storrow AB, Wu AH, Christenson RH, Apple FS, Francis G, Tang W; National Academy of Clinical Biochemistry. National Academy of Clinical Biochemistry Laboratory Medicine Practice Guidelines: clinical characteristics and utilization of biochemical markers in acute coronary syndromes. Clin Chem. 2007 Apr;53(4):552-74. doi: 10.1373/clinchem.2006.084194. Epub 2007 Mar 23. No abstract available. PMID 17384001
- [Result] Wang TK, Stewart RA, Ramanathan T, Kang N, Gamble G, White HD. Diagnosis of MI after CABG with high-sensitivity troponin T and new ECG or echocardiogram changes: relationship with mortality and validation of the universal definition of MI. Eur Heart J Acute Cardiovasc Care. 2013 Dec;2(4):323-33. doi: 10.1177/2048872613496941. Epub 2013 Aug 5. PMID 24338291
- [Result] Lurati Buse GA, Koller MT, Grapow M, Bolliger D, Seeberger M, Filipovic M. The prognostic value of troponin release after adult cardiac surgery - a meta-analysis. Eur J Cardiothorac Surg. 2010 Feb;37(2):399-406. doi: 10.1016/j.ejcts.2009.05.054. Epub 2009 Aug 20. PMID 19699102
- [Result] Apple FS, Jesse RL, Newby LK, Wu AH, Christenson RH; National Academy of Clinical Biochemistry; IFCC Committee for Standardization of Markers of Cardiac Damage. National Academy of Clinical Biochemistry and IFCC Committee for Standardization of Markers of Cardiac Damage Laboratory Medicine Practice Guidelines: Analytical issues for biochemical markers of acute coronary syndromes. Circulation. 2007 Apr 3;115(13):e352-5. doi: 10.1161/CIRCULATIONAHA.107.182881. Epub 2007 Mar 23. No abstract available. PMID 17384332
- [Result] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Writing Group on behalf of the Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of Myocardial Infarction. Third universal definition of myocardial infarction. Glob Heart. 2012 Dec;7(4):275-95. doi: 10.1016/j.gheart.2012.08.001. Epub 2012 Sep 26. No abstract available. PMID 25689940